CLINICAL TRIAL: NCT03957382
Title: Evaluation of Safety and Efficacy of the Accero® (Heal) Stent for Intracranial Aneurysm Treatment
Status: Active, not recruiting | Type: Observational
Sponsor: Acandis GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: 1041-1
Record Dates: First submitted 2019-05-16; First posted 2019-05-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Stents

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Accero® (heal) Stent — The Accero® (heal) Stent will only be used in line with the Instructions For Use (IFU). Patients participating in this PMCF (Post- Market Clinical Follow-up) will not be exposed to any additional risk. There are no additional treatments or investigations other than done in the clinical routine.

SUMMARY:
This study is intended to show that the application of the Accero® (heal) stent is safe within the given indication.

ELIGIBILITY:
Inclusion Criteria:

Any patient treated with ACCERO® (heal) Stent according to IFU and has signed the informed consent

Exclusion Criteria:

- Patient is participating in another clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients treated with Accero® (heal) Stent
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2019-07-23 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Raymond Roy Classification | 6 months after treatment
  Assessment of Raymond Roy Classification
Raymond Roy Classification | 12 months after treatment
  Assessment of Raymond Roy Classification
Raymond Roy Classification | 24 months after treatment
  Assessment of Raymond Roy Classification
Raymond Roy Classification | 36 months after treatment
  Assessment of Raymond Roy Classification

SECONDARY OUTCOMES:
modified Rankin Scale (mRS) | 6 months after treatment
  Assessment of modified Rankin Scale
  Modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities.
  The scale runs from 0-6:
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
modified Rankin Scale (mRS) | 12 months after treatment
  Assessment of modified Rankin Scale
  Modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities.
  The scale runs from 0-6:
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
modified Rankin Scale (mRS) | 24 months after treatment
  Assessment of modified Rankin Scale
  Modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities.
  The scale runs from 0-6:
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
modified Rankin Scale (mRS) | 36 months after treatment
  Assessment of modified Rankin Scale
  Modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities.
  The scale runs from 0-6:
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.

CONTACTS AND LOCATIONS:
Overall Officials: Maxim Bester, PD. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (4):
- Germany (4):
  - Klinik und Poliklinik für Neuroradiologische Diagnostik und Intervention, Universitätsklinikum Hamburg-Eppendorf, Hamburg, Hamburg
  - Vivantes - Klinikum Neukölln Institut für klinische und interventionelle Neuroradiologie, Berlin
  - Krankenhaus Ludmillenstift, Abteilung für Radiologie, Neuroradiologie und Nuklearmedizin, Meppen
  - KLINIKUM VEST GMBH Knappschaftskrankenhaus Klinik für Radiologie und Neuroradiologie, Recklinghausen

IPD SHARING:
Plan to Share IPD: No